CLINICAL TRIAL: NCT06756087
Title: Radiofrequency Ablation/Vertebroplasty Versus Radiofrequency Ablation/Vertebroplasty Combined with SBRT for Painful Spinal Vertebral Metastases: a Multicenter, Practical, Randomized, Controlled, Non-Inferiority Clinical Study
Brief Title: Evaluate the Efficacy of Radiofrequency Ablation/Vertebroplasty with or Without SBRT for Treating Painful Spinal Vertebral Metastases
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: The Third Affiliated Hospital of Southern Medical University (Other Government); Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Dongqing Zuo, Principal Investigator, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20240912033813578
Record Dates: First submitted 2024-12-16; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-11

CONDITIONS: Spinal Metastases; Local Control; Pain Cancer
Keywords: spinal metastases; Radiofrequency Ablation; Stereotactic radiotherapy
MeSH Terms: conditions — Cancer Pain | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Radiofrequency ablation/vertebroplasty (Experimental): Patients underwent OsteoCool radiofrequency ablation and vertebroplasty for spinal metastatic tumors. After the operation, the original anti-tumor treatment was continued within 1-2 weeks according to the recovery. Local intervention was no longer carried out at the operation site, and the normal follow-up was started.
  Interventions: Radiation: Radiofrequency Ablation (RFA)/Vertebroplasty+Stereotactic Radiotherapy
- Standard control: Ablation/Vertebroplasty and SBRT Radiotherapy (Other): Patients underwent OsteoCool radiofrequency ablation and vertebroplastyfor spinal metastatic tumors. Then were sent to SBRT radiotherapy 2-3 weeks postoperatively. follow-up visit start at the end of adiotherapy.
  Interventions: Procedure: Experimental

INTERVENTIONS:
Radiation: Radiofrequency Ablation (RFA)/Vertebroplasty+Stereotactic Radiotherapy — All patients received OsteoCool™ radiofrequency ablation + vertebroplasty for spinal metastatic tumors at the Department of Bone Oncology, Shanghai First People's Hospital.
  Standard Control Group: Patients received SBRT (Stereotactic Body Radiation Therapy) from the Department of Radiation Oncology 2-3 weeks post-surgery. This included pre-radiation positioning, mold preparation, and radiation therapy. After radiation therapy, patients rested for 2 weeks before resuming their original anti-tumor treatment and starting follow-up.SBRT therapy was administered according to the recommendations, using one of the following dose and fractionation schemes: 4 sessions of 24 Gy, 5 sessions of 30 Gy, 6 sessions of 36 Gy, or 7 sessions of 42 Gy.
  Arms: Radiofrequency ablation/vertebroplasty
Procedure: Experimental — patients received OsteoCool™ radiofrequency ablation+vertebroplasty for spinal metastatic tumors at the Department of Bone Oncology, Shanghai First People's Hospital. patients continued their original anti-tumor treatment within 1-2 weeks based on their recovery. No further local intervention was performed at the surgical site, and normal follow-up was started.
  Arms: Standard control: Ablation/Vertebroplasty and SBRT Radiotherapy

SUMMARY:
This study is a prospective, multicenter, open, practical, randomized controlled, non inferiority effect clinical study initiated by researchers, which aims to evaluate the clinical efficacy and safety of radiofrequency ablation/vertebroplasty and radiofrequency ablation/vertebroplasty combined with SBRT in the treatment of painful spinal metastases. This study plans to include about 120 cases in about 3 research centers nationwide, including the Department of bone oncology of Shanghai First People's Hospital (main center, 60 cases), the Department of bone oncology of the Third Affiliated Hospital of Southern Medical University (sub center 1, 30 cases), and the Department of bone oncology of Peking University People's Hospital (sub center 2, 30 cases). The patient was diagnosed with spinal metastasis of malignant tumor and had pain of more than 3 points. The subjects with spinal metastasis located at t5-l5 were selected for clinical research. All patients were treated with RFA/PVA minimally invasive surgery. In principle, no more than 2 vertebral bodies were treated. All patients will receive MRI/CT examination of the affected spine within 6 weeks before enrollment to determine the degree of spinal involvement. All patients were randomly divided into experimental group and control group after minimally invasive surgery, the ratio was 1:1. The patients in the experimental group recovered to the original system treatment about two weeks after minimally invasive surgery; The control group began to receive SBRT radiotherapy of the surgical vertebral body in about two weeks, and the radiotherapy time was two weeks. According to the recommendations of the Department of radiotherapy, SBRT radiotherapy should use any of the following dose and grading scheme: 4 times 24gy, 5 times 30Gy, 6 times 36Gy, 7 times 42GY. The patients in the two groups were followed up after treatment, and evaluated at 1, 2 and 4 weeks and 3, 6 and 12 months after treatment. The NRPS pain degree and pafi pain function comprehensive score were evaluated, and the local lesions were evaluated at 1, 3, 6 and 12 months after operation. To evaluate the local control of spinal metastases, pain improvement and quality of life changes of the two treatment strategies.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, open, practical, randomized controlled, non inferiority effect clinical study initiated by researchers, which aims to evaluate the clinical efficacy and safety of radiofrequency ablation/vertebroplasty and radiofrequency ablation/vertebroplasty combined with SBRT in the treatment of painful spinal metastases. This study plans to include about 120 cases in about 3 research centers nationwide, including the Department of bone oncology of Shanghai First People's Hospital (main center, 60 cases), the Department of bone oncology of the Third Affiliated Hospital of Southern Medical University (sub center 1, 30 cases), and the Department of bone oncology of Peking University People's Hospital (sub center 2, 30 cases). The patient was diagnosed with spinal metastasis of malignant tumor and had pain of more than 3 points. The subjects with spinal metastasis located at t5-l5 were selected for clinical research. All patients were treated with RFA/PVA minimally invasive surgery. In principle, no more than 2 vertebral bodies were treated. All patients will receive MRI/CT examination of the affected spine within 6 weeks before enrollment to determine the degree of spinal involvement. All patients were randomly divided into experimental group and control group after minimally invasive surgery, the ratio was 1:1. The patients in the experimental group recovered to the original system treatment about two weeks after minimally invasive surgery; The control group began to receive SBRT radiotherapy of the surgical vertebral body in about two weeks, and the radiotherapy time was two weeks. According to the recommendations of the Department of radiotherapy, SBRT radiotherapy should use any of the following dose and grading scheme: 4 times 24gy, 5 times 30Gy, 6 times 36Gy, 7 times 42GY. The patients in the two groups were followed up after treatment, and evaluated at 1, 2 and 4 weeks and 3, 6 and 12 months after treatment. The NRPS pain degree and pafi pain function comprehensive score were evaluated, and the local lesions were evaluated at 1, 3, 6 and 12 months after operation. To evaluate the local control of spinal metastases, pain improvement and quality of life changes of the two treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

1. The subject voluntarily participates in this study, and both the patient and their family sign an informed consent form. The subject demonstrates good compliance and cooperates with follow-up.
2. Age 18 or older, no gender restrictions.
3. The target population for this trial consists of patients with bone metastases from malignant tumors confirmed by pathology or imaging, with lesions located between T5 and L5. The number of affected vertebral sites is fewer than three, and the lesions are mainly osteolytic, affecting primarily the vertebral bodies.
4. Expected survival is greater than three months.
5. Initial diagnosis with an NPRS pain score > 3.
6. ECOG performance status score of 0-2.
7. The function of vital organs meets the following requirements: a) Adequate bone marrow function: WBC ≥ 3.0×10^9/L; absolute neutrophil count (ANC) ≥ 1.5 ×10^9/L; lymphocyte count ≥ 6.0×10^8/L; platelet count ≥ 50×10^9/L, with no blood transfusion within 14 days prior to the first cellular therapy; hemoglobin ≥ 10.0 g/dL. b) Adequate liver and kidney function: total bilirubin ≤ 2.0×ULN, AST and ALT < 2.5×ULN; serum creatinine ≤ 1.5×ULN, or creatinine clearance ≥ 50 ml/min (calculated using the Cockcroft-Gault formula). c) Coagulation function: INR ≤ 1.5×ULN, APTT ≤ 1.5×ULN. d) Adequate cardiovascular function: left ventricular ejection fraction (EF) ≥ 50%, QTcF interval ≤ 450 ms for males and ≤ 470 ms for females.
8. Use of at least one medically approved contraceptive method (e.g., surgical sterilization, oral contraceptives, intrauterine device, abstinence, or barrier methods with spermicide) for at least six months.

Exclusion Criteria:

1. Subjects with no measurable lesions;
2. Known brain metastasis and/or clinically suspected brain metastasis (subjects with asymptomatic brain metastasis or clinically stable brain metastasis for more than three months after local treatment can be included);
3. Subjects whose target lesions received radiotherapy within the past two years;
4. Tumor types sensitive to radiotherapy, including malignant lymphoma, testicular seminoma, Wilms tumor, neuroblastoma, medulloblastoma, Ewing sarcoma, and small cell tumors.
5. Spinal metastases involving spinal appendages, destruction of the posterior wall of the vertebral canal, or compression of the spinal dura mater;
6. Subjects preparing for or who have previously undergone tissue/organ transplantation;
7. Subjects with active infections or unexplained fever >38.5℃ during screening or before treatment;
8. Patients with active pulmonary tuberculosis (TB), currently receiving anti-TB treatment or treated for TB within the past year before screening;
9. Positive syphilis serology test;
10. Known history of HIV-positive test or known acquired immunodeficiency syndrome (AIDS);
11. Active hepatitis B: hepatitis B surface antigen (HBsAg) positive with HBV DNA levels exceeding 10,000 IU/ml; hepatitis C: hepatitis C antibody (HCV Ab) positive with HCV RNA levels exceeding 1,000 IU/ml; co-infection with hepatitis B and hepatitis C;
12. Cardiovascular disease meeting any of the following: a. Congestive heart failure with NYHA classification ≥ III; b. Severe arrhythmia requiring medication; c. Acute myocardial infarction, severe or unstable angina, coronary or peripheral artery bypass grafting, or stenting within six months before initial dosing; d. Left ventricular ejection fraction (LVEF) < 50%; e. QTcF interval > 450 ms for males and > 470 ms for females, or risk factors for torsades de pointes, such as clinically significant hypokalemia, family history of long QT syndrome, or familial arrhythmias (e.g., Wolff-Parkinson-White syndrome) as determined by the investigator;
13. Uncontrolled hypertension (defined as systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg despite standardized antihypertensive treatment);
14. Subjects deemed by the investigator to have serious uncontrolled diseases or other conditions that may affect participation in the study or render them unsuitable for study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male or female not limited.
Enrollment: 120 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Compare the pain control of RFA/PVA and RFA/PVA combined with SBRT radiotherapy for painful spinal metastases. | 1, 2, and 4 weeks after treatment, as well as at 3, 6, and 12 months
  Based on NRPS pain score: Compare the pain scores of two groups of patients at 1, 2, and 4 weeks after treatment, as well as at 3, 6, and 12 months after treatment.
  The Numerical Pain Rating (NPR) Scale is used to assess the intensity of a patient's pain. The pain intensity is rated using numbers from 0 to 10, where 0 represents no pain, and 10 represents the most intense pain imaginable. The patient is asked to select a number that best represents their level of pain, or a healthcare provider may assist in understanding the scale and help the patient choose the appropriate number to describe their pain.
  Based on the pain score, pain severity is classified as follows:
  Mild pain (1-3): Does not affect sleep. Moderate pain (4-6): Affects sleep. Severe pain (7-10): Significantly disrupts sleep. During the course of treatment, patients are expected to take pain medication as needed. Pain assessments should be performed 20 minutes before the patient takes their pain medication each day.

SECONDARY OUTCOMES:
Comparison of local control between RFA/PVA and RFA/PVA combined with SBRT radiotherapy for painful spinal metastases | 1, 3, 6, and 12 months after treatment
  Evaluate and calculate the DCR of local lesions in two groups of patients at 1, 3, 6, and 12 months after treatment based on the MDA bone response standard.
  DCR (Disease Control Rate) refers to the proportion of patients with spinal metastatic tumors who achieve the best therapeutic response according to the The MDA Bone Response Criteria (MD Anderson Bone Response Criteria) is a set of imaging-based criteria used to assess the treatment response in patients with bone metastatic tumors. The criteria are typically applied in clinical trials and research studies to evaluate the effect of various treatments (such as chemotherapy.MDA bone response criteria, as assessed by imaging. This includes patients who achieve Complete Response (CR), Partial Response (PR), or Stable Disease (SD) after treatment.
  All patients undergo CT or MRI scans at the designated follow-up time points. The imaging measurements and assessments are performed by the same physician (HJ) who evaluates the results.
Compare the limb function of RFA/PVA and RFA/PVA combined with SBRT radiotherapy in the treatment of painful spinal metastases; | 1, 3, 6, and 12 months after treatment.
  Based on the Combined Pain and Ambulatory Function Index, calculate the comprehensive PAFI pain function of two groups of patients at 1, 3, 6, and 12 months after treatment.
  Combined Pain and Ambulatory Function Index and Evaluation Time
  10 points - Normal walking and recreational activities: No pain or limp. 9 points - Normal walking ability: Mild pain but no limp; no need for walking aids (crutches, cane, walker).
  8 points - Walking ability: Moderate pain and mild limp; rarely uses (or prefers not to use) walking aids (crutches, cane, walker).
  7 points - Walking ability with walking aids: Severe pain while walking without walking aids; mild pain when using walking aids (crutches, cane, walker).
  6 points - Walking ability with walking aids: Moderate pain when using walking aids (crutches, cane, walker).
  5 points - Walking with walking aids: Severe pain and significant limping when using walking aids (crutches, cane, walker).
  4 points - Unable to walk, using a wheelchair: Can sit in

CONTACTS AND LOCATIONS:
Overall Officials: Dongqing Zuo, M.D./PH.D., Study Director — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
1. Ethical Concerns Participant Confidentiality: Even with de-identification, there is a risk that participants could be re-identified, especially in small or unique populations.
     Consent Limitations: Participants may not have explicitly consented to sharing their data for secondary use or may have only agreed to specific types of research.
  2. Risk of Misuse Misinterpretation of Data: Secondary users might misinterpret the data due to a lack of context or understanding of the study.
  Data Misuse: There is a risk that the data could be used for purposes that contradict the original intent of the research or that harm participants or specific groups.